CLINICAL TRIAL: NCT02631343
Title: A Community-based Model of Delivery of Kangaroo Mother Care for Improving Child Survival and Brain Development in Low Birth Weight Newborns
Brief Title: Community Kangaroo Mother Care for Improving Child Survival and Brain Development in Low Birth Weight Newborns
Acronym: CKMC-DEV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Society for Applied Studies (Other)
Collaborators: Grand Challenges Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0725-03
Record Dates: First submitted 2015-11-25; First posted 2015-12-16 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Low Birth Weight
Keywords: Kangaroo mother care in the community

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention KMC (Experimental): Promotion of, and support for lactation management and skin to skin care as soon as possible after birth by study ANM supported by study ASHA in addition to routine visits by government health workers
  Interventions: Behavioral: KMC; Other: Essential newborn care
- Control (Other): Routine visits by government health workers
  Interventions: Other: Essential newborn care

INTERVENTIONS:
Behavioral: KMC — Promotion of, and support for lactation management and skin to skin care as soon as possible after birth by study ANM supported by study ASHA in addition to routine visits by government health workers
  Arms: Intervention KMC
Other: Essential newborn care

SUMMARY:
While newborn and child survival remains a priority, optimal development of survivors is receiving increasing attention. Interventions that impact both survival and development should be prioritized for action. Kangaroo Mother Care (KMC) improves survival, and potentially neurodevelopment, in preterm and low birth weight infants in hospital settings but its coverage remains low. Innovation is required to allow the community-based delivery of KMC by front-line workers. This could greatly accelerate scale up and sustainability of this intervention in low resource settings.

The proposed randomized trial is planned in a setting where 40% of births take place at home. Early discharge (as early as within 12 hours of birth) is common for facility births, often at the request of families for social and cultural reasons. Many of the hospitals do not have incubators for the care of very small babies.

DETAILED DESCRIPTION:
Low birth weight (LBW) infants will be identified through surveillance. Eligible infants will be randomized into the intervention and control groups. Mother in the intervention group will be supported by a ANM-like study workers assisted by ASHA-like study workers to provide Kangaroo mother care (KMC) to their babies at home. Breastfeeding support will also be provided to these mothers by ANM-like study workers. Essential newborn care will be delivered through Government workers in both groups. Survival will be measured in all enrolled infants through contacts at 1, 3, 6 and 12 months of age. Information will also be ascertained on initiation of breastfeeding, exclusive breastfeeding rates, incidence of infection in the neonatal and in the 1-5 months period. Development outcomes (Maternal Depression, Maternal sense of competence, Mother-infant Bonding, Mother-infant interaction, Newborn Behaviour, Infant temperament, Brain development) will be measured at enrolment, 6weeks, 6 and 12 months of age. Growth will be measured at enrolment and at 1, 3, 6 and 12 months.

ELIGIBILITY:
Inclusion criteria

- Mothers and low birth weight ≥1500gms to ≤2250gms

Exclusion criteria

* Birth weight <1500gms
* Unable to feed on offering feeds, confirmed by study team
* Infant has breathing problems or less active
* Mother does not intend to stay in study area for the next 12 months

Max Age: 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 550 (Actual)
Dates: Start 2015-11; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Assessment of maternal depression | 6 weeks
  The depression will be measured using patient health questionnaire-9
Assessment of maternal depression | Assessment of maternal depression at 6 months
  The depression will be measured using patient health questionnaire-9
Assessment of maternal sense of competence | 6 weeks
  Maternal sense of competence will be measured by maternal self efficacy questionnaire
Assessment of maternal sense of competence | Assessment of maternal sense of competence at 12 months
  Maternal sense of competence will be measured by maternal self efficacy questionnaire
Assessment of mother infant bonding | 6 weeks
  Mother infant bonding will be measured by maternal postnatal attachment questionnaire
Assessment of mother infant interaction | 6 months
  Mother infant interaction will be assessed by video recording and subsequent coding of Joint attention task
Assessment of newborn behaviour | 6 weeks
  Assessment of newborn behaviour by Neonatal behavioural assessment scale
Assessment of infant temperament | 6 months
  Assessment of infant temperament by infant temperament scale
Assessment of infant temperament | Assessment of infant temperament at 12 months
  Assessment of infant temperament by infant temperament scale
Assessment of cognitive function by Bayley scale | 6 months
Assessment of cognitive function by Bayley scale | Assessment of cognitive function by Bayley scale at 12 months
Assessment of home environment by PROCESS | 12 months

SECONDARY OUTCOMES:
Neonatal mortality | From birth to 28 days
Early infant mortality | From birth to 6 months
Early initiation of breastfeeding | From birth to 1 month
Proportion exclusively breastfed | 1, 3 and 6 months
Weight and length gain | 1, 3, 6 and 12 months
Incidence of infection in neonatal | 1 month period
Early recognition of illness at 1 month | 1 month period
  Recognition of illness and careseeking will be ascertained from caregivers by using questionnaires
Early and appropriate care seeking practices at 1 month | 1 month period
  Early and appropriate care seeking ascertained from caregivers by using questionnaires
Early recognition of illness at 3 months | Assessed at 3 months data from 1 month upto 3 months
Early and appropriate care seeking practices at 3 months | Assessed at 3 months data from 1 month upto 3 months
Early recognition of illness at 6 months | Assessed at 6 months data from 3 months upto 6 months
Early and appropriate care seeking practices at 6 months | Assessed at 6 months data from 3 months upto 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sunita Taneja, MBBS, PhD, Principal Investigator — Centre for Health Research and Development, Society for Applied Studies
Locations (1):
- CHRD, Society for Applied Studies, Palwal, Haryana, India

REFERENCES:
- [Derived] Upadhyay RP, Taneja S, Strand TA, Sommerfelt H, Hysing M, Mazumder S, Bhandari N, Martines J, Dua T, Kariger P, Bahl R. Early child stimulation, linear growth and neurodevelopment in low birth weight infants. BMC Pediatr. 2022 Oct 8;22(1):586. doi: 10.1186/s12887-022-03579-6. PMID 36209050
- [Derived] Taneja S, Sinha B, Upadhyay RP, Mazumder S, Sommerfelt H, Martines J, Dalpath SK, Gupta R, Kariger P, Bahl R, Bhandari N, Dua T; ciKMC development study group. Community initiated kangaroo mother care and early child development in low birth weight infants in India-a randomized controlled trial. BMC Pediatr. 2020 Apr 4;20(1):150. doi: 10.1186/s12887-020-02046-4. PMID 32247311
- [Derived] Mazumder S, Taneja S, Dube B, Bhatia K, Ghosh R, Shekhar M, Sinha B, Bahl R, Martines J, Bhan MK, Sommerfelt H, Bhandari N. Effect of community-initiated kangaroo mother care on survival of infants with low birthweight: a randomised controlled trial. Lancet. 2019 Nov 9;394(10210):1724-1736. doi: 10.1016/S0140-6736(19)32223-8. Epub 2019 Oct 4. PMID 31590989